CLINICAL TRIAL: NCT04561037
Title: Efficacy of Adding Pulsed Electromagnetic Field Therapy to Mobilization and Exercises in Patients With TMJ Dysfunction After Facial Penetrating Injury: Randomized Single-blinded Study
Brief Title: Pulsed Electromagnetic Field Therapy for TMJ Dysfunction After Facial Penetrating Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Kadry, Lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control group patients received traditional physical therapy treatment. The traditional physical therapy treatment program consisted of TMJ mobilization techniques include distraction, anterior glide, anterior glide with pre-positioned mouth opening, medial/lateral glides, caudal-anterior-medial (CAM) glide, and CAM glide with pre-positioned mouth opening and isometric exercises against resistance for muscles of mastication.
  Interventions: Other: TMJ physical therapy program
- Study Group (Experimental): Study group patients received PEMFT, using EMG 8400 PEMF device (made in Italy, by EME) in addition to physical therapy treatment program.
  Interventions: Device: Pulsed Electromagnetic Field therapy (PEMFT)

INTERVENTIONS:
Device: Pulsed Electromagnetic Field therapy (PEMFT) — PEMFT was connected to electrical mains supplying 220v. Pair of applicators sized 16x10x3 cm was adjust to be over TMJ, on both sides of the face; the appliance was adjusted to the frequency of 50 HZ and intensity of 90 Gauss. Twelve PEMF treatment sessions of 30 min duration were provided 3 times per week TMJ mobilization techniques and isometric exercises against resistance for muscles of mastication
  Arms: Study Group
Other: TMJ physical therapy program — TMJ manual physical therapy program (mobilization and gentle isometric exercises) for 30, 3 times a week, for 4 weeks.
  Arms: Control Group

SUMMARY:
This study is aiming to investigate the effect of magnetic therapy in combination with traditional physical therapy on the pain and mouth opening, after facial penetrating wound injury with no facial fractures, that treated conservatively

ELIGIBILITY:
Inclusion Criteria:

* TMJ pain and mouth opening limitation after 1 month of facial penetrating wound injury as the wound is fully healed.
* TMJ pain (in 1 or both joints) after facial penetrating wound injury.

Exclusion Criteria:

* Patient excluded from the study if they had one of the following:
* TMJ fracture or dislocation
* Previous TMJ surgeries
* Dental diseases
* Infectious or systemic diseases
* Pregnancy
* Malignancy
* Pacemaker or metal implants
* Systemic diseases that affect joint function such as rheumatoid arthritis.

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in the Maximum mouth opening in millimeter (mm) before and after intervention. | Change between baseline and 4 weeks of treatment measures.
  Each participant was asked to open his or her mouth as wide as possible after that the examiner used a digital Vernier caliper to measure the maximum vertical distance from the incisal edge of the upper central incisors to the incisal edge of the lower central incisors at the midline

SECONDARY OUTCOMES:
Change in TMJ pain measured by Visual Analogue Scale (VAS) | Change between baseline and 4 weeks of treatment measures.
  Visual Analogue Scale (VAS) was used to evaluate pain intensity. VAS is a subjective pain measurement method consisting of a straight line of 100 mm on which patients scored their pain intensity where 0 corresponds to no pain and 10 corresponds to the worst maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kadry, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers upon request and after discussion with the research team